CLINICAL TRIAL: NCT05565105
Title: A Phase II Trial of CD34+ Enriched Transplants From HLA-Compatible Related or Unrelated Donors for Treatment of Patients With Leukemia or Lymphoma
Brief Title: CD34+ Transplants for Leukemia and Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guenther Koehne (Other)
Responsible Party: Sponsor-Investigator, Guenther Koehne, Deputy Director and Chief of Blood and Marrow Transplant, Hematologic Oncology and Benign Hematology, Baptist Health South Florida
Organization: Baptist Health South Florida (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KOE-001
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Acute
Keywords: Stem Cell Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Whole-Body Irradiation; Thiotepa; Cyclophosphamide; Busulfan; Melphalan; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Regimen A: TBI/Thiotepa/Cyclophosphamide (Experimental): Patients in enrolled in Regimen A will receive the following:
  * Total Body Irradiation (TBI), hyper-fractionated to a dose of 1320 cGy depending on age, stage of disease and requirement of general anesthesia with lung shielding
  * Thiotepa, 5 mg/kg/day x 2 days via IV infusion over 4 hours daily or 10 mg/kg on one day
  * Cyclophosphamide, 60 mg/kg/day x 2 days via IV infusion over 2 hours daily (or if cyclophosphamide is contraindicated, fludarabine at 25 mg/m^2 x 5 days may be substituted)
  Interventions: Radiation: Total Body Irradiation (TBI); Drug: Thiotepa; Drug: Cyclophosphamide
- Regimen B: Busulfan/Melphalan/Fludarabine (Experimental): Patients in enrolled in Regimen B will receive the following:
  * Busulfan, IV 0.8 mg/kg q6hours x 10 or 12 doses over 3 days, depending on the disease
  * Melphalan, 70 mg/m^2/day x 2 days via IV infusion over 30 minutes daily
  * Fludarabine, 25 mg/m^2/day x 5 days via IV infusion over 30 minutes daily
  Interventions: Drug: Busulfan; Drug: Melphalan; Drug: Fludarabine

INTERVENTIONS:
Radiation: Total Body Irradiation (TBI) — Hyper-fractioned TBI is administered by a linear accelerator at a dose rate of < 15 cGy/minute.
  Arms: Regimen A: TBI/Thiotepa/Cyclophosphamide
Drug: Thiotepa — Thiotepa: 5 mg/kg/day IV over approximately 4 hours daily x 2 (Day -5 and Day -4).
  Other Names: Thioplex
  Arms: Regimen A: TBI/Thiotepa/Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide: 60 mg/kg/day x 2 or Fludarabine 25 mg/m^2 x 5 if cyclophosphamide is contraindicated
  Other Names: Cytoxan
  Arms: Regimen A: TBI/Thiotepa/Cyclophosphamide
Drug: Busulfan — Busulfan: 0.8 mg/kg every 6 hours x 10 or 12 doses (depending on disease) with dose modified according to pharmacokinetics
  Other Names: Busulfex
  Arms: Regimen B: Busulfan/Melphalan/Fludarabine
Drug: Melphalan — Melphalan: 70 mg/m^2/day x 2
  Other Names: Alkeran
  Arms: Regimen B: Busulfan/Melphalan/Fludarabine
Drug: Fludarabine — Fludarabine: 25 mg/m^2/day x 5
  Other Names: Fludara
  Arms: Regimen B: Busulfan/Melphalan/Fludarabine

SUMMARY:
This study will evaluate whether processing blood stem cell transplants using an investigational device (the CliniMACS system) results in less complications for patients undergoing transplant for treatment of a blood malignancy (cancer) or blood disorder.

ELIGIBILITY:
Inclusion Criteria:

* Malignant conditions or other life-threatening disorders correctable by transplant for which CD34+ selected, T-cell depleted allogeneic hematopoietic stem cell transplantation is indicated such as:

  1. AML in 1st remission - for patients who is AML does not have 'good risk' cytogenetic features (i.e. t8:21, t 15: 17, inv16).
  2. Secondary AML in 1st remission
  3. AML in 1st relapse or 2nd remission
  4. ALL/CLL in patient remission clinical or molecular features indicating a high risk for relapse; or ALL/CLL 2nd remission
  5. CML failing to respond to or not tolerating imatinib or dasatinib in first chronic phase of disease; CML in accelerated phase, second chronic phase, or in CR after accelerated phase or blast crisis.
  6. Non-Hodgkin's lymphoma with chemo responsive disease in any of the following categories:

     1. Intermediate or high-grade lymphomas who have failed to achieve a first CR or have relapsed following a 1st remission who are not candidates for autologous transplants.
     2. Any NHL in remission which is considered not curable with chemotherapy alone and not eligible/appropriate for autologous transplant.
  7. Chronic myelomonocyte leukemia: CMML-1 and CMML-2.

The following inclusion criteria are also required:

* Patient's age includes from ≥18 to ≤74 years old.
* Patients may be of either gender or any ethnic background.
* Patients must have a Karnofsky (adult) Performance Status of at least 70%
* Patients must have adequate organ function measured by:

Cardiac: asymptomatic or if symptomatic then LVEF at rest must be 50% and must improve with exercise.

Hepatic: < 3x ULN AST and: s 1.5 total serum bilirubin, unless there is congenital benign hyperbilirubinemia or if the hyperbilirubinemia is directly caused by the disease in which the patient is receiving a transplant (e.g. AML Chloroma obstructing the biliary tree). Patients with higher bilirubin levels due to causes other than active liver disease is also eligible with Pl approval e.g. patients with PNH, Gilbert's disease or other hemolytic disorders.

Renal: serum creatinine: s; 1.2 mg/dL or if serum creatinine is outside the normal range, then CrCl > 30 ml/min (measured or calculated/estimated).

Pulmonary: asymptomatic or if symptomatic, DLCO 50% of predicted (corrected for hemoglobin).

Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Patient seropositive for HIV-I /II; HTLV -I /II
* Presence of leukemia in the CNS

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of graft versus host disease (GvHD) | Two years
  Incidence of acute and chronic GvHD
Severity of disease | Two years
  Severity of the adverse events will be reported based on the CTCAE Version 5.
Incidence of transplant-related mortality (TRM) | Two years
  TRM includes fatal complications resulting from the allogeneic transplant and/ or treatment regimens such as graft failure, GvHD, hemorrhages, and infections.
Change in overall survival (OS) | Six months, one year, two years
  OS is defined as time from transplant to death or last follow-up.
Change in disease free survival (DFS) | Six months, one year, two years
  DFS is defined as the minimum time interval of times to relapse/recurrence, to death or to the last follow- up, from the time of transplant.

SECONDARY OUTCOMES:
Proportion of patients optimal and suboptimal doses | Two years
  The proportion of patients receiving optimal cell doses (CD34+: >5x 10^6/kg and CD3+: < 5 x10^4/kg) and suboptimal doses (CD34+: <3 x 10^6/kg and CD3+: >5 x 10^4/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Guenther Koehne, MD, PhD, Principal Investigator — Baptist Health South Florida/Miami Cancer Institute
Locations (1):
- Baptist Health South Florida/Miami Cancer Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Handgretinger R, Klingebiel T, Lang P, Schumm M, Neu S, Geiselhart A, Bader P, Schlegel PG, Greil J, Stachel D, Herzog RJ, Niethammer D. Megadose transplantation of purified peripheral blood CD34(+) progenitor cells from HLA-mismatched parental donors in children. Bone Marrow Transplant. 2001 Apr;27(8):777-83. doi: 10.1038/sj.bmt.1702996. PMID 11477433
- [Background] Urbano-Ispizua A, Rozman C, Pimentel P, Solano C, de la Rubia J, Brunet S, Perez-Oteyza J, Ferra C, Zuazu J, Caballero D, Bargay J, Carvalhais A, Diez JL, Espigado I, Alegre A, Rovira M, Campilho F, Odriozola J, Sanz MA, Sierra J, Garcia-Conde J, Montserrat E; Spanish Group for Allogeneic Peripheral Blood Transplantation (Grupo Espanol de Trasplante Hemopoyetico) and Instituto Portugues de Oncologia-Porto. Risk factors for acute graft-versus-host disease in patients undergoing transplantation with CD34+ selected blood cells from HLA-identical siblings. Blood. 2002 Jul 15;100(2):724-7. doi: 10.1182/blood-2001-11-0057. PMID 12091376
- [Background] Jakubowski AA, Small TN, Young JW, Kernan NA, Castro-Malaspina H, Hsu KC, Perales MA, Collins N, Cisek C, Chiu M, van den Brink MR, O'Reilly RJ, Papadopoulos EB. T cell depleted stem-cell transplantation for adults with hematologic malignancies: sustained engraftment of HLA-matched related donor grafts without the use of antithymocyte globulin. Blood. 2007 Dec 15;110(13):4552-9. doi: 10.1182/blood-2007-06-093880. Epub 2007 Aug 23. PMID 17717135
- See also: Miami Cancer Institute — https://baptisthealth.net/services/cancer-care/miami-cancer-institute